CLINICAL TRIAL: NCT00768560
Title: Evaluation of the Efficacy, Safety, and Pharmacokinetics/Pharmacodynamics of BAY A1040 CR Tablet on High Dose Administration in Patients With Essential Hypertension.
Brief Title: Nifedipine (Adalat CR, BAY A1040) High Dose PK/PD Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13012
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nifedipine; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nifedipine (Adalat CR, BAYA1040) 40 mg OD (Active Comparator): Nifedipine (Adalat CR, BAYA1040) 40 milligram (mg) once daily (OD) in the morning
  Interventions: Drug: Nifedipine (Adalat CR, BAYA1040) 40mg OD
- Nifedipine (Adalat CR, BAYA1040) 40 mg BID (Experimental): Nifedipine (Adalat CR, BAYA1040) 40 milligram (mg) twice daily (BID). 40 mg in the morning and 40 mg in the evening
  Interventions: Drug: Nifedipine (Adalat CR, BAYA1040) 40mg BID
- Nifedipine (Adalat CR, BAYA1040) 80 mg OD (Experimental): Nifedipine (Adalat CR, BAYA1040) 80 milligram (mg) once daily (OD) in the morning
  Interventions: Drug: Nifedipine (Adalat CR, BAYA1040) 80mg OD

INTERVENTIONS:
Drug: Nifedipine (Adalat CR, BAYA1040) 80mg OD — Nifedipine (Adalat CR, BAYA1040) 80 milligram (mg) once daily (OD) in the morning
  Arms: Nifedipine (Adalat CR, BAYA1040) 80 mg OD
Drug: Nifedipine (Adalat CR, BAYA1040) 40mg BID — Nifedipine (Adalat CR, BAYA1040) 40 milligram (mg) twice daily (BID). 40 mg in the morning and 40 mg in the evening
  Arms: Nifedipine (Adalat CR, BAYA1040) 40 mg BID
Drug: Nifedipine (Adalat CR, BAYA1040) 40mg OD — Nifedipine (Adalat CR, BAYA1040) 40 milligram (mg) once daily (OD) in the morning
  Arms: Nifedipine (Adalat CR, BAYA1040) 40 mg OD

SUMMARY:
This is a multi-center, randomized, double-blind, 6 x 3 cross-over study. All patients who meet the entry criteria will be required to stop taking any other anti-hypertensive agents than Adalat CR (controlled release), if taken, before starting 4 weeks (±7days) open-label Adalat CR 40 mg once daily (OD) treatment phase (baseline treatment period). Of them, those who are confirmed with their eligibility as subjects for the present study at the end of the baseline treatment period will be randomly allocated to one of the 6 treatment sequences on the basis of a computer-generated randomization list. Subsequently, BAY A1040 CR tablet 40 mg OD, 40 mg twice daily (BID) or 80 mg OD will be administered to a total of 6 weeks, 2 weeks per each treatment period (Period 1-3) under double-blind conditions using BAY A1040 CR tablet 40 mg and its placebo as follows (Double-blind treatment period).

DETAILED DESCRIPTION:
Issues on safety are addressed in the Adverse Event section.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* 20 years or older and less than 75 years
* Outpatient
* Untreated or treated patients with antihypertensive agents whose blood pressure (BP) in sitting position at entry (Visit 1) is as follows.

  * Untreated patients: systolic blood pressure (SBP) >= 160mmHg or diastolic blood pressure (DBP) >= 100mmHg
  * Treated patients: SBP >= 140mmHg or DBP >= 90mmHg (at trough)

Exclusion Criteria:

* Patients whose BP during baseline treatment period is: SBP>=200mmHg or DBP>=120mmHg.
* Patients with secondary hypertension or hypertensive emergency.
* Patients with cardiovascular or cerebrovascular ischemic event (stroke, transient ischemic attack (TIA), myocardial infarction or unstable angina), or with history of these within 6 months prior to the study.
* Patients with intracranial or subarachnoid hemorrhage, or with history of these within 6 months prior to the study.
* Patients with server hematopoietic dysfunction (acute/chronic leukemia, myeloma, malignant lymphoma, myelodysplastic syndrome, aplastic anemia), or with history of these.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Japan (3):
  - Sendai, Miyagi
  - Suita, Osaka
  - Koshigaya, Saitama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 47 subjects were recruited from 30 Jan 2008 to 11 May 2008 by 3 centers in Japan.
Pre-assignment Details: After a 4-week baseline treatment with Adalat controlled release (CR) 40 mg once daily (OD), 35 subjects were randomized to double-blind treatment and were included in the safety analysis. 34 subjects were included in the analysis of pharmacokinetics, efficacy and demographic data. 1 subject discontinued the study in Period 1 due to adverse event.
Period: Intervention Set 1
Arm/Group | Nifedipine 40 mg OD x 40 mg BID x 80 mg OD for 2 Weeks Each | Nifedipine 40 mg OD x 80 mg OD x 40 mg BID for 2 Weeks Each | Nifedipine 40 mg BID x 80 mg OD x 40 mg OD for 2 Weeks Each | Nifedipine 40 mg BID x 40 mg OD x 80 mg OD for 2 Weeks Each | Nifedipine 80 mg OD x 40 mg OD x 40 mg BID for 2 Weeks Each | Nifedipine 80 mg OD x 40 mg BID x 40 mg OD for 2 Weeks Each
Started | 5 (3-period/treatment crossover) | 6 (3-period/treatment crossover) | 6 (3-period/treatment crossover) | 6 (3-period/treatment crossover) | 6 (3-period/treatment crossover) | 6 (3-period/treatment crossover)
Subjects Received Treatment | 5 (40 mg OD for 2 weeks) | 6 (40 mg OD for 2 weeks) | 6 (40 mg twice daily (BID) for 2 weeks) | 6 (40 mg BID for 2 weeks) | 6 (80 mg OD for 2 weeks) | 6 (80 mg OD for 2 weeks)
Completed | 5 | 5 | 6 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Intervention Set 2
Arm/Group | Nifedipine 40 mg OD x 40 mg BID x 80 mg OD for 2 Weeks Each | Nifedipine 40 mg OD x 80 mg OD x 40 mg BID for 2 Weeks Each | Nifedipine 40 mg BID x 80 mg OD x 40 mg OD for 2 Weeks Each | Nifedipine 40 mg BID x 40 mg OD x 80 mg OD for 2 Weeks Each | Nifedipine 80 mg OD x 40 mg OD x 40 mg BID for 2 Weeks Each | Nifedipine 80 mg OD x 40 mg BID x 40 mg OD for 2 Weeks Each
Started | 5 (40 mg BID for 2 weeks) | 5 (80 mg OD for 2 weeks) | 6 (80 mg OD for 2 weeks) | 6 (40 mg OD for 2 weeks) | 6 (40 mg OD for 2 weeks) | 6 (40 mg BID for 2 weeks)
Completed | 5 | 5 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Set 3
Arm/Group | Nifedipine 40 mg OD x 40 mg BID x 80 mg OD for 2 Weeks Each | Nifedipine 40 mg OD x 80 mg OD x 40 mg BID for 2 Weeks Each | Nifedipine 40 mg BID x 80 mg OD x 40 mg OD for 2 Weeks Each | Nifedipine 40 mg BID x 40 mg OD x 80 mg OD for 2 Weeks Each | Nifedipine 80 mg OD x 40 mg OD x 40 mg BID for 2 Weeks Each | Nifedipine 80 mg OD x 40 mg BID x 40 mg OD for 2 Weeks Each
Started | 5 (80 mg OD for 2 weeks) | 5 (40 mg BID for 2 weeks) | 6 (40 mg OD for 2 weeks) | 6 (80 mg OD for 2 weeks) | 6 (40 mg BID for 2 weeks) | 6 (40 mg OD for 2 weeks)
Completed | 5 | 5 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nifedipine 40 mg OD x 40 mg BID x 80 mg OD for 2 Weeks Each | Nifedipine 40 mg OD x 80 mg OD x 40 mg BID for 2 Weeks Each | Nifedipine 40 mg BID x 80 mg OD x 40 mg OD for 2 Weeks Each | Nifedipine 40 mg BID x 40 mg OD x 80 mg OD for 2 Weeks Each | Nifedipine 80 mg OD x 40 mg OD x 40 mg BID for 2 Weeks Each | Nifedipine 80 mg OD x 40 mg BID x 40 mg OD for 2 Weeks Each | Total
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 34
Age, Continuous [Mean (Full Range); unit: years] | 61.4 [55 to 68] | 63.6 [55 to 73] | 59.7 [55 to 65] | 64.3 [60 to 70] | 58.2 [37 to 67] | 59.7 [56 to 68] | 61.1 [37 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 2 | 1 | 1 | 8
  Male | 4 | 2 | 6 | 4 | 5 | 5 | 26
Blood Pressure (Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)) at Baseline [Mean (Standard Deviation); unit: mm Hg] — Blood pressure (BP) before the start of baseline treatment. Subjects valid for safety analysis
  mm Hg
    SBP at baseline | 150.00 (7.91) | 161.00 (16.67) | 156.33 (11.18) | 155.83 (10.96) | 156.33 (14.79) | 154.83 (13.53) | 155.89 (12.38)
    DBP at baseline | 94.40 (4.98) | 95.00 (6.60) | 98.00 (6.45) | 91.00 (7.07) | 92.50 (3.45) | 89.83 (7.68) | 93.43 (6.40)
Heart rate (HR) at Baseline [Mean (Standard Deviation); unit: beats / min] — Heart rate (HR) before the start of baseline treatment. Subjects valid for safety analysis
  beats / min | 64.20 (6.18) | 72.67 (13.95) | 79.00 (10.81) | 70.83 (5.42) | 68.50 (7.87) | 79.50 (17.84) | 72.69 (11.83)

OUTCOME MEASURES:

1. Primary Outcome: Change of Sitting Blood Pressure
Description: Changes of sitting SBP and DBP (trough values) from baseline (ie [trough BP at the end of each period during the double-blind treatment period] minus [trough BP at the end of the baseline treatment period])
Time Frame: Baseline and after 2 weeks treatment
Population: Per-protocol efficacy population: subjects valid for safety analysis who have no critical protocol deviation and have trough BP at the end of baseline treatment period and trough BP at the end of period 1 are considered valid for the analysis.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Nifedipine (Adalat CR, BAYA1040) 40 mg OD | Nifedipine (Adalat CR, BAYA1040) 40 mg BID | Nifedipine (Adalat CR, BAYA1040) 80 mg OD
Number analyzed (Participants) | 34 | 34 | 34
mm Hg
  Systolic Blood Pressure | -10.19 (1.24) | -19.88 (1.24) | -10.13 (1.24)
  Diastolic Blood Pressure | -4.30 (0.65) | -8.28 (0.65) | -4.98 (0.65)
Statistical Analysis 1: Comparison: Nifedipine (Adalat CR, BAYA1040) 40 mg OD vs Nifedipine (Adalat CR, BAYA1040) 40 mg BID; The point estimate and 90% confidence interval of the difference of changes in SBP from baseline was estimated by using the analysis of variance (ANOVA) model including the terms: group, subject within a group, dosage and administration and stage as fixed effects; Test type: Superiority or Other; Mean Difference (Final Values) = -9.69, 90% CI [-12.62 to -6.77] — 40 mg BID minus 40 mg OD
Statistical Analysis 2: Comparison: Nifedipine (Adalat CR, BAYA1040) 40 mg OD vs Nifedipine (Adalat CR, BAYA1040) 80 mg OD; The point estimate and 90% confidence interval of the difference of changes in SBP from baseline was estimated by using the ANOVA model including the terms: group, subject within a group, dosage and administration and stage as fixed effects; Test type: Superiority or Other; Mean Difference (Final Values) = 0.06, 90% CI [-2.87 to 2.98] — 80 mg OD minus 40 mg OD
Statistical Analysis 3: Comparison: Nifedipine (Adalat CR, BAYA1040) 40 mg BID vs Nifedipine (Adalat CR, BAYA1040) 80 mg OD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Mean Difference (Final Values) = 9.75, 90% CI [6.83 to 12.67] — 80 mg OD minus 40 mg BID
Statistical Analysis 4: Comparison: Nifedipine (Adalat CR, BAYA1040) 40 mg OD vs Nifedipine (Adalat CR, BAYA1040) 40 mg BID; The point estimate and 90% confidence interval of the difference of changes in DBP from baseline was estimated by using the ANOVA model including the terms: group, subject within a group, dosage and administration and stage as fixed effects; Test type: Superiority or Other; Mean Difference (Final Values) = -3.97, 90% CI [-5.50 to -2.44] — 40 mg BID minus 40 mg OD
Statistical Analysis 5: Comparison: Nifedipine (Adalat CR, BAYA1040) 40 mg OD vs Nifedipine (Adalat CR, BAYA1040) 80 mg OD; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.68, 90% CI [-2.21 to 0.85] — 80 mg OD minus 40 mg OD
Statistical Analysis 6: Comparison: Nifedipine (Adalat CR, BAYA1040) 40 mg BID vs Nifedipine (Adalat CR, BAYA1040) 80 mg OD; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.29, 90% CI [1.76 to 4.82] — 80 mg OD minus 40 mg BID

2. Secondary Outcome: Differences of Systolic Blood Pressure Profile
Description: Differences in blood pressure at the same time points (0, 2, 4, 6, 8, 10, 12, 24-hour post-dose) between 2 different days (ie, end of baseline treatment period and end of 2-week treatment period)
Time Frame: Baseline and after 2 weeks treatment
Population: Subjects valid for efficacy analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nifedipine (Adalat CR, BAYA1040) 40 mg OD | Nifedipine (Adalat CR, BAYA1040) 40 mg BID | Nifedipine (Adalat CR, BAYA1040) 80 mg OD
Number analyzed (Participants) | 34 | 34 | 34
mm Hg
  At 0-hour post-dose | -11.35 (15.75) | -21.24 (11.56) | -9.91 (10.58)
  At 2-hour post-dose | -4.91 (11.62) | -8.65 (11.19) | -11.97 (10.15)
  At 4-hour post-dose | -6.18 (12.05) | -5.76 (11.25) | -7.85 (10.02)
  At 6-hour post-dose | -6.56 (12.58) | -4.94 (9.31) | -7.26 (8.40)
  At 8-hour post-dose | -7.88 (11.53) | -6.97 (10.23) | -7.88 (10.68)
  At 10-hour post-dose | -4.79 (10.60) | -4.03 (10.64) | -6.56 (9.41)
  At 12-hour post-dose | -5.59 (10.98) | -4.38 (9.31) | -6.00 (9.98)
  At 24-hour post-dose | -8.97 (12.79) | -18.38 (8.34) | -10.21 (10.87)

3. Secondary Outcome: Differences of Diastolic Blood Pressure Profile
Description: as for outcome 2
Time Frame: Baseline and after 2 weeks treatment
Population: Subjects valid for efficacy analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nifedipine (Adalat CR, BAYA1040) 40 mg OD | Nifedipine (Adalat CR, BAYA1040) 40 mg BID | Nifedipine (Adalat CR, BAYA1040) 80 mg OD
Number analyzed (Participants) | 34 | 34 | 34
mm Hg
  At 0-hour post-dose | -3.82 (6.40) | -8.12 (6.24) | -4.18 (5.54)
  At 2-hour post-dose | -4.15 (7.27) | -5.47 (7.01) | -7.18 (5.89)
  At 4-hour post dose | -3.44 (7.47) | -1.62 (8.11) | -3.68 (6.33)
  At 6-hour post-dose | -5.56 (7.42) | -1.71 (7.20) | -3.85 (5.94)
  At 8-hour post dose | -3.09 (6.13) | -3.18 (6.26) | -4.74 (6.30)
  At 10-hour post-dose | -2.24 (6.34) | -1.74 (6.42) | -3.82 (7.26)
  At 12-hour post-dose | -2.47 (6.59) | -2.15 (7.30) | -3.15 (6.97)
  At 24-hour post dose | -5.00 (7.34) | -8.47 (5.39) | -5.82 (8.18)

4. Secondary Outcome: Target Blood Pressure Achievement in Elderly (≥65)
Description: Elderly subjects (≥65 years) without diabetes mellitus or chronic renal disorders and target BP SBP <140 mm Hg and DBP <90 mm Hg
Time Frame: After 2 weeks treatment
Population: Subjects valid for efficacy analysis
Measure: Number; unit: participants
Arm/Group | Nifedipine (Adalat CR, BAYA1040) 40 mg OD | Nifedipine (Adalat CR, BAYA1040) 40 mg BID | Nifedipine (Adalat CR, BAYA1040) 80 mg OD
Number analyzed (Participants) | 5 | 5 | 5
participants | 2 | 3 | 3

5. Secondary Outcome: Target Blood Pressure Achievement in Non-elderly (<65)
Description: Non-elderly subjects (<65 years) without diabetes mellitus or chronic renal disorder and target BP SBP <130 mm Hg and DBP <85 mm Hg
Time Frame: After 2 weeks treatment
Population: Subjects valid for efficacy analysis
Measure: Number; unit: participants
Arm/Group | Nifedipine (Adalat CR, BAYA1040) 40 mg OD | Nifedipine (Adalat CR, BAYA1040) 40 mg BID | Nifedipine (Adalat CR, BAYA1040) 80 mg OD
Number analyzed (Participants) | 14 | 14 | 14
participants | 3 | 10 | 4

6. Secondary Outcome: Target Blood Pressure Achievement in Subjects With Diabetes Mellitus or Chronic Renal Disorder
Description: Subjects with diabetes mellitus or chronic renal disorders and target BP SBP <130 mm Hg and DBP <80 mm Hg
Time Frame: After 2 weeks treatment
Population: Subjects valid for efficacy analysis
Measure: Number; unit: participants
Arm/Group | Nifedipine (Adalat CR, BAYA1040) 40 mg OD | Nifedipine (Adalat CR, BAYA1040) 40 mg BID | Nifedipine (Adalat CR, BAYA1040) 80 mg OD
Number analyzed (Participants) | 15 | 15 | 15
participants | 0 | 4 | 1

7. Secondary Outcome: Target Blood Pressure Achievement in All Subjects
Description: Subjects (≥65 years) without diabetes mellitus or chronic renal disorders and target BP SBP <140 mm Hg and DBP <90 mm Hg. Subjects (<65 years) without diabetes mellitus or chronic renal disorder and target BP SBP <130 mm Hg and DBP <85 mm Hg. Subjects with diabetes mellitus or chronic renal disorders and target BP SBP <130 mm Hg and DBP <80 mm Hg.
Time Frame: After 2 weeks treatment
Population: Subjects valid for efficacy analysis
Measure: Number; unit: participants
Arm/Group | Nifedipine (Adalat CR, BAYA1040) 40 mg OD | Nifedipine (Adalat CR, BAYA1040) 40 mg BID | Nifedipine (Adalat CR, BAYA1040) 80 mg OD
Number analyzed (Participants) | 34 | 34 | 34
participants | 5 | 17 | 8

ADVERSE EVENTS:
Arm/Group | Nifedipine (Adalat CR, BAYA1040) 40 mg OD | Nifedipine (Adalat CR, BAYA1040) 40 mg BID | Nifedipine (Adalat CR, BAYA1040) 80 mg OD
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 5/35 | 7/34 | 5/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nifedipine (Adalat CR, BAYA1040) 40 mg OD (N=35) | Nifedipine (Adalat CR, BAYA1040) 40 mg BID (N=34) | Nifedipine (Adalat CR, BAYA1040) 80 mg OD (N=34)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Blood albumin decreased (Investigations) | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Cardiac murmur (Cardiac disorders) | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1
Lipid metabolism disorder (Metabolism and nutrition disorders) | 1 | 1 | 0
Carotid arteriosclerosis (Cardiac disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less